CLINICAL TRIAL: NCT02040116
Title: Study Evaluating Rapid Infusion Rituximab in Patients With Autoimmune Diseases
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00022197
Record Dates: First submitted 2014-01-14; First posted 2014-01-20 (Estimated); Results first posted 2017-09-20 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-08

CONDITIONS: Multiple Sclerosis
Keywords: Rapid Infusion Rituximab
MeSH Terms: conditions — Multiple Sclerosis | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- rituximab infusion (Other): Every patient is getting the same therapy of rituximab. If day 1 is tolerated at standard infusion then day 14 and beyond will be given as rapid infusion over 90 minutes
  Interventions: Drug: Rituximab Infusion

INTERVENTIONS:
Drug: Rituximab Infusion — Participants will receive their first infusion of rituximab at the standard infusion rate provided in the manufacturer labeling. If they tolerate this infusion with a grade 2 of less infusion-related reaction, the next infusion will be administered as a 90 minute rapid infusion.
  Other Names: Rituxan

SUMMARY:
The purpose of this study is to evaluate the impact of rapid infusion rituximab on the incidence of infusion-related reactions in patients with Autoimmune Diseases.

DETAILED DESCRIPTION:
Background Rituximab is a human/murine monoclonal antibody targeted at the CD20 antigen (cluster of differentiation antigen 20) on B-lymphocytes. The CD20 antigen is expressed in over 90% of B-cell non-Hodgkin's lymphomas. B cells are also believed to play a role in the pathogenesis of other oncologic and non-oncologic disorders. Targeting B cells appears to have a role in decreasing autoimmune and inflammatory processes, as well as antibody production in many autoimmune diseases. Rituximab is approved for the treatment of non-Hodgkin's lymphoma (NHL), chronic lymphocytic leukemia (CLL), rheumatoid arthritis (RA) in combination with methotrexate, wegener's granulomatosis, and microscopic polyangiitis in combination with glucocorticoids. Although rituximab is not approved for multiple sclerosis, myasthenia gravis, or other autoimmune diseases, it is commonly used later in the treatment course for patients that are not responding to other treatment options. Rituximab's main limitation is the occurrence of infusion-related reactions (IRR). These reactions can include fever, chills, rash, respiratory compromise, and a variety of other symptoms, including death. The incidence of IRR is known to vary depending on the rituximab indication. The incidence of IRR with the first infusion of rituximab is approximately 77% with NHL, 27% with RA, and 12% with wegener's granulomatosis and microscopic polyangiitis. The incidence of IRR decreases with subsequent infusions of rituximab to approximately 5-10%. According to the National Cancer Institute, there are 5 grades of IRR. In general, grade 1 reactions are classified as asymptomatic or only mild symptoms that do not require intervention. Grade 2 reactions are classified as moderate with minimal, local, or noninvasive interventions required. Grade 3 reactions are classified as severe and medically significant, but not immediately life-threatening. These reactions require hospitalization or prolongation of a current hospitalization. Grade 4 reactions are classified as life-threatening with urgent interventions required. Grade 5 reactions are classified as death related to an adverse drug event. The incidence of IRR is a chief concern for patients, nurses, and other healthcare providers.

The package labeling recommends the administration of a standard infusion of rituximab for all patients initiating rituximab therapy to minimize IRR. If this infusion is tolerated then subsequent infusions may be titrated up to a faster rate to decrease infusion time. Based on the manufacturer's package insert, rituximab is infused at a rate of 50 mg/hr and can be increased every 30 minutes by 50 mg/hr (maximum rate of 400 mg/hr). If a grade 3 or 4 IRR does not occur, subsequent infusions are given at a rate of 100 mg/hr and can be increased every 30 minutes by 100 mg/hr (maximum rate of 400 mg/hr). The average infusion time is estimated to be 4-6 hours for the first infusion, and 3-4 hours for subsequent infusions. Rituximab is typically given in cycles and the timing will vary depending on the indication.

ELIGIBILITY:
Inclusion Criteria:

* Autoimmune patient at Wake Forest Baptist Health that is eligible for rituximab therapy
* Tolerate the standard infusion rituximab with ≤ grade 2 hypersensitivity reaction
* Consent to participate in the rapid infusion study
* Age ≥ 18 years ≤ 80 years

Exclusion Criteria:

* Tolerate the standard infusion rituximab with ≥ grade 3 hypersensitivity reaction
* Neurocognitive impairment (i.e. dementia, Alzheimers, et al)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: LeAnne D Kennedy, PharmD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab Infusion: Every patient is getting the same therapy of rituximab. If day 1 is tolerated at standard infusion then day 14 and beyond will be given as rapid infusion over 90 minutes
  Rapid Infusion Rituximab: Participants will receive their first infusion of rituximab at the standard infusion rate provided in the manufacturer labeling. If they tolerate this infusion with a grade 2 of less infusion-related reaction, the next infusion will be administered as a 90 minute rapid infusion.
Period: Overall Study
Arm/Group | Rituximab Infusion
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Rituximab Infusion: Every patient is getting the same therapy of rituximab. If day 1 is tolerated at standard infusion then day 14 and beyond will be given as rapid infusion over 20 hours
  Rapid Infusion Rituximab: Participants will receive their first infusion of rituximab at the standard infusion rate provided in the manufacturer labeling. If they tolerate this infusion with a grade 2 of less infusion-related reaction, the next infusion will be administered as a 90 minute rapid infusion.
Arm/Group | Rituximab Infusion
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 40 [30 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Infusion Related Reactions With Rapid Infusion Will be Reported
Description: Patients are given therapy on day 1 and if infusion is tolerated with < grade 2 reaction based on the CTCAE v4 then then will proceed to rapid infusion on day 14 which is given over 90 minutes. The number of infusion reaction is measured for all patients and in all infusions given.
Time Frame: 14 Days
Measure: Number; unit: infusion reactions
Groups:
- Number of Reactions for Standard Infusion: day 1 infusion of standard infusion will be given the same to all patients and then assessed
- Number of Reactions for Rapid Infusion: day 1 infusion of rapid infusion will be given the same to all patients and then assessed
Arm/Group | Number of Reactions for Standard Infusion | Number of Reactions for Rapid Infusion
Number analyzed (Participants) | 19 | 19
infusion reactions | 0 | 0

2. Secondary Outcome: Change in Chair Time With Rapid Infusion Will be Reported
Description: The amount of time spent administering the rituximab will be compared to the time from the first infusion to the second infusion. The change was calculated from two time points as the value at the later time point minus the value at the earlier time point.
Time Frame: 14 Days
Measure: Mean (Full Range); unit: Hours
Groups:
- Time in Day Hospital: The time of infusion will be recorded from the first dose and the second dose
  Time in day hospital: time between the two doses will recorded
Arm/Group | Time in Day Hospital
Number analyzed (Participants) | 19
Hours | -10 [-21 to -1]

3. Primary Outcome: Grade of Infusion Related Reactions With Rapid Infusion Will be Reported
Description: Patients are given therapy on day 1 and if infusion is tolerated with < grade 2 reaction based on the CTCAE v4 then then will proceed to rapid infusion on day 14 which is given over 90 minutes. The grade of infusion reaction is measured for all patients and in all infusions given. According to the National Cancer Institute, there are 5 grades of IRR. In general, grade 1 reactions are classified as asymptomatic or only mild symptoms that do not require intervention. Grade 2 reactions are classified as moderate with minimal, local, or noninvasive interventions required. Grade 3 reactions are classified as severe and medically significant, but not immediately life-threatening. These reactions require hospitalization or prolongation of a current hospitalization. Grade 4 reactions are classified as life-threatening with urgent interventions required. Grade 5 reactions are classified as death related to an adverse drug event.
Time Frame: 14 Days
Population: Due to their being no reactions, the Grade of reactions for Standard infusion will and can not be reported, as the lowest grade requires there to be a reaction.
Groups:
- Grade of Reactions for Standard Infusion: day 1 infusion of standard infusion will be graded according to CTCAE
- Grade of Reactions for Rapid Infusion: day 14 infusion of standard infusion will be graded according to CTCAE
Arm/Group | Grade of Reactions for Standard Infusion | Grade of Reactions for Rapid Infusion
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Rituximab Infusion
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No